CLINICAL TRIAL: NCT07160738
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, TWO-COHORT, TWO-PERIOD, FIXED SEQUENCE STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSES OF ITRACONAZOLE AND PROBENECID ON THE PHARMACOKINETICS OF SINGLE DOSE PF-07220060 ADMINISTERED UNDER THE FED CONDITION TO HEALTHY PARTICIPANTS
Brief Title: A Study to Learn About How the Study Medicines Called Itraconazole and Probenecid Change How the Body Processes PF-07220060
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C4391011
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults
Keywords: probenecid; breast cancer; CDK4 inhibitor; itraconazole; PF-07220060; Drug-Drug Interaction (DDI)
MeSH Terms: conditions — Breast Neoplasms | interventions — Itraconazole; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Period 1: PF-07220060 (Experimental): In Cohort 1, Period 1 participants will receive a single dose of PF-07220060 tablet given orally and administered with food on Day 1.
  Interventions: Drug: PF-07220060
- Cohort 1, Period 2: PF-07220060 and itraconazole (Experimental): In Cohort 1 Period 2, participants will receive oral dose of itraconazole once daily from Day 1 to Day 9. On the morning of Day 4, participants will first receive one oral dose of itraconazole followed by a single oral dose of PF-07220060 tablet
  Interventions: Drug: PF-07220060; Drug: Itraconazole
- Cohort 2, Period 1: PF-07220060 (Experimental): In Cohort 2, Period 1 participants will receive a single dose of PF-07220060 tablet given orally and administered with food on Day 1.
  Interventions: Drug: PF-07220060
- Cohort 2, Period 2: PF-07220060 probenecid (Experimental): In Cohort 2, Period 2, participants will receive oral dose of probenecid four times a day from Day 1 to Day 9. On the morning of Day 3, participants will first receive one oral dose of probenecid followed by a single oral dose of PF-07220060 tablet.
  Interventions: Drug: PF-07220060; Drug: Probenecid

INTERVENTIONS:
Drug: PF-07220060 — Tablet given orally
Drug: Itraconazole — Capsule given orally
  Arms: Cohort 1, Period 2: PF-07220060 and itraconazole
Drug: Probenecid — Tablet given orally
  Arms: Cohort 2, Period 2: PF-07220060 probenecid

SUMMARY:
The purpose of the study is to see and learn the effect of multiple doses of a strong CYP3A4 inhibitor and a potent UGT2B7 inhibitor on the PK of PF-07220060.

DETAILED DESCRIPTION:
This study is seeking participants who are:

1. male and female aged 18 to 65 years and are healthy as confirmed by medical tests 2. with body mass index (BMI) of 17.5-30.5 kilogram per meter squared (kg/m2); and a total body weight of more than 50 kilograms (110 pounds).

The study will consist of 2 groups each containing 2 periods. In both groups, participants will receive a single dose of PF-07220060 in Period 1. In group 1 Period 2, itraconazole will be given once a day from Day 1 to Day 9. On the morning of Period 2 Day 4, a single dose of PF 07220060 will be taken by mouth immediately after itraconazole is taken by mouth. In group 2 Period 2, probenecid will be given 4 times a day from Day 1 to Day 9. On the morning of Period 2 Day 3, a single dose of PF 07220060 will be taken by mouth, immediately after probenecid is taken by mouth.

In both groups, PF-07220060 will be given by mouth about 30 minutes after a moderate fat standard calorie meal in Period 1. In cohort 1 Period 2, itraconazole will be given by mouth once a day from Day 1 to Day 9 about 30 minutes after a moderate fat standard calorie meal. On the morning of Period 2 Day 4, a single dose of PF 07220060 will be administered by mouth immediately after itraconazole administration. In cohort 2 Period 2, probenecid will be given by mouth 4 times a day (QID) with 6±2 hours intervals from Day 1 to Day 9 with or without food. On Period 2 Day 2, the last probenecid dose prior to the Day 3 first dose will be given under fasted condition. On the morning of Period 2 Day 3, after 10 hours fasting, ~30 min after a moderate fat standard calorie breakfast, a single dose of PF-07220060 will be administered by mouth, immediately after probenecid administration.

The study will look at the effect of multiple doses of itraconazole and probenecid on how the body processes a single oral dose of PF-07220060.

Participants will take part in this study for up to 78 days for group 1 and 77 days for group 2. Following period 1 and 2, they will undergo lab tests and blood samples will be collected after administration of PF-07220060. Participants will be discharged from the research unit at the end of period 2 following completion of all tests.

ELIGIBILITY:
Inclusion

* Healthy volunteers who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
* Body mass index (BMI) of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated Informed Consent Document (ICD) indicating that the participant has been informed of all pertinent aspects of the study.

Exclusion

* Evidence or history of blood dyscrasias, uric acid kidney stones, peptic ulcer or gout for probenecid cohort (Applicable to Cohort 2).
* Evidence or history of genetic deficiency of glucose -6- phosphate dehydrogenase in red blood cells for probenecid cohort (Applicable to Cohort 2).
* Concomitant use of any medications or substances that are strong inducers or inhibitors of CYP3A4 or UGT2B7 are prohibited within 5 half-lives plus 14 days (up to 28 days) prior to first dose of PF 07220060.
* Concomitant use of methotrexate, salicylates, penicillin or other beta-lactams, sulfonamide, ketamine, thiopental anesthesia, indomethacin, naproxen, ketoprofen, meclofenamate, lorazepam are prohibited within 5 half-lives plus 14 days (up to 28 days) prior to first dose of PF 07220060 (Applicable to Cohort 2).
* History of sensitivity to azole antifungals, probenecid, or any of the formulation components of PF-07220060.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-01-09 (Estimated)

PRIMARY OUTCOMES:
Plasma PF-07220060 Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post PF-07220060 dose for Period 1; Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post PF-07220060 dose for Period 2
Plasma PF-07220060 Area under the plasma concentration versus time curve (AUC) | Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post PF-07220060 dose for Period 1; Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours post PF-07220060 dose for Period 2

SECONDARY OUTCOMES:
Number of Participants With Laboratory Abnormalities | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Treatment-Emergent Adverse Events (AEs) | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | From baseline up to 28 to 35 days after last dose of investigational drug
Number of participants taking concomitant medications | From baseline up to 28 to 35 days after last dose of investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391011